CLINICAL TRIAL: NCT00234559
Title: A Randomized Controlled Study Comparing Vacuum Assisted Closure® Therapy to Moist Wound Therapy in Angiogenesis
Brief Title: Trial of Vacuum Assisted Closure® Therapy Versus Control Therapy in Angiogenesis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to no subject enrollment.
Sponsor: KCI USA, Inc (Industry)
Organization: Solventum US LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VACP2005-001
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Wounds
Keywords: Angiogenesis; Post surgical dehisced wounds of the lower extremity
MeSH Terms: conditions — Wounds and Injuries

INTERVENTIONS:
Device: VAC® Therapy System

SUMMARY:
The purpose of this study is to determine:

1. If vacuum assisted closure (VAC®) therapy results in altered proteomic expression of angiogenic markers compared to moist wound therapy.
2. If VAC® therapy results in increased angiogenesis compared to moist wound therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female and > 18 years old.
* Patient or patient's legal authorized representative is willing to sign informed consent.
* Patient has a post surgical dehisced wound of the lower extremity for longer than two weeks and less than one month.
* Patient has transcutaneous oximetry (TcPO2) evaluation that demonstrated tissue hypoxia in the periwound region, as indicated by a reading of 10-40 mmHg within the prior two weeks.
* Ankle Brachial Index > 0.7 within the prior two weeks.
* Patient is not pregnant (pregnancy test is negative) and non-lactating at Visit 1.
* Patient does not plan on becoming pregnant during the course of the study.
* Patient is willing to use effective method of contraception for the duration of the study, is permanently sterilized, or post-menopausal as defined by cessation of menses for at least one year prior to enrollment in study.

Exclusion Criteria:

* Diagnosed and untreated wound infection.
* Poor nutrition status as evidenced by pre-albumin < 12mg/dl within the past 30 days or extracellular mass < 95%.
* Presence of sickle cell disease.
* Presence of connective tissue disease (e.g. history of or active lupus).
* Hemoglobin A1c (HbA1c) levels greater than 9% thirty days prior to screening visit (if patient is confirmed diabetic).
* Treatment with an investigational therapy within the previous 30 days.
* Lower extremity wound (under consideration for study) with malignancy.
* Lower extremity wound (under consideration for study) with untreatable cellulitis.
* Presence of untreated osteomyelitis.
* Presence of any systemic hematologic disorder or condition that would impede healing.
* History of radiation to the wound area.
* History of drugs that may delay wound healing.
* History of thermal injury to the wound area.
* Prior VAC® therapy to the wound within 30 days of enrollment.
* Current or prior treatment with hyperbaric oxygen therapy (HBO) or warm-up therapy to the same wound.
* Recent diagnosis of cancer or active management of cancer within the last year.
* Treatment with skin or dermal substitutes or dressings with living cells capable of producing growth factors within the previous 30 days.
* End stage renal disease.
* History of alcohol or drug abuse that may impact protocol compliance or delay wound healing.
* Known hypersensitivity to hydrogel or any disposable component of the VAC® Therapy System.
* Necrotic tissue with eschar present which cannot be debrided.
* Any other severe concurrent disease, which, in the judgment of the investigator, would make the patient inappropriate for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Altered proteomic expression evaluated by angiogenic markers using biomolecular assays of biopsy samples at Day 0, Day 3, Day 7, Day 21, and Day 28

SECONDARY OUTCOMES:
Increased angiogenesis of the lower extremity wound will be quantified using the MicroScan™ (video microscope) at Day 0, Day 3, Day 7, Day 21, Day 28, Day 42, and at follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Niezgoda, M.D., Principal Investigator — St. Luke's Medical Center of Aurora Health Care